CLINICAL TRIAL: NCT07281742
Title: Amblyopia Treatment for Children Aged 8 to 12 Years
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 2024-0924
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Amblyopia
Keywords: amblyopia; dichoptic; children
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with Curesight videos (Experimental): with this IRB application), indicated for improvement in visual acuity and stereo acuity in amblyopia patients, aged 4 - <9 years, associated with anisometropia and/or with mild strabismus. This approval was based on data from a pilot study and a multi-center randomized clinical trial conducted with children aged 4 to 8 years.25,26 However, very few children older than age 7 years were included so the effectiveness of Curesight™ treatment for children aged 8 to 12 is unknown. Our pilot study will evaluate response to the Curesight™ treatment in this older age range.
  Interventions: Device: Curesight dichoptic videos

INTERVENTIONS:
Device: Curesight dichoptic videos — Streamed videos are converted into 2 anaglyph channels, blue images for the amblyopic eye and red images for the fellow eye, and are presented superimposed. The stronger eye has blur imposed in the central visual area; the weaker amblyopic eye channel is not affected by the blur.

SUMMARY:
This study is being done to assess the effect of at-home amblyopia treatment with Curesight™ for children aged 8 to 12 years. Curesight™ allows you to stream any videos on a computer screen at home but the amblyopic eye will see the entire screen clearly while part of the image will be blurred for the other eye. There is already a pivotal clinical trial showing that this treatment is effective for young children and Curesight™ has been cleared for use as an amblyopia treatment by the FDA for children as young as 4 years.

DETAILED DESCRIPTION:
Amblyopia (lazy eye) is a developmental vision disorder in which the brain doesn't efficiently process images from one eye and which over time causes decreased vision in that eye. Early detection and early treatment, by age 7 years, are effective in reducing the burden of amblyopia. There is evidence from randomized clinical trials (RCTs) that 73-90% of amblyopic children in this age range treated with glasses and patching, the most commonly prescribed treatments for amblyopia, have improvements in visual acuity. More recently, binocular amblyopia treatments show similar effectiveness to patching in children <7 years old. Yet, full recovery of normal visual acuity occurs in only 30-40% of children regardless of treatment approach; most amblyopic children have residual amblyopia post-treatment at age 8-12 years, when there is little or no benefit of additional or other standard-of care treatments. It is important investigate novel treatments for amblyopia in older children because the vision deficits in persistent residual amblyopia also have associated knock-on effects, including slow reading and impaired motor skills in natural binocular viewing conditions, diminished self-perception and reduced quality of life. Failure to detect and remediate amblyopia during childhood typically results in lifelong deficits and doubles the lifelong risk of visual impairment in the fellow eye.

To address this need, we will conduct a pilot study to investigate whether the novel Curesight™ is effective in treating amblyopia in older children aged 8 to 12 years. CureSight™ is an eye-tracking based system designed to treat amblyopia under dichoptic conditions that incorporates eye-tracking and separation of streamed visual stimuli presented on a tablet into 2 separate digital channels, one for each eye . The treatment task consists of passively watching streamed video content presented by the system according to the child's personal preference from the web links approved by the parents. The main components of the system include : (1) a an 11.6-inch tablet for viewing the videos (2) an eye tracker bar placed below the tablet that tracks each eye's gaze position, (3) anaglyph (red-cyan) glasses worn while watching videos to separate stimuli presented to each eye and (4) proprietary software that uses the eye-tracking data to blur the central vision area of the visual stimuli presented to the fellow eye to encourage the brain to use the sharp, high resolution information from the amblyopic eye's center of vision. The diameter and magnitude of the blur are adjusted automatically during treatment according to the visual of each eye, as measured at follow-up visits, entered on the CureSight™ cloud portal (Health Insurance Portability and Accountability Act and General Data Protection Regulation compliant). Worse amblyopic eye visual acuity and larger differences in visual acuity between eyes result in more blur and greater diameter of blur. The Curesight™ device received Food and Drug Administration clearance (identifier, K221375; September 29, 2022; uploaded with this IRB application), indicated for improvement in visual acuity and stereo acuity in amblyopia patients, aged 4 - <9 years, associated with anisometropia and/or with mild strabismus. This approval was based on data from a pilot study and a multi-center randomized clinical trial conducted with children aged 4 to 8 years.25,26 However, very few children older than age 7 years were included so the effectiveness of Curesight™ treatment for children aged 8 to 12 is unknown. Our pilot study will evaluate response to the Curesight™ treatment in this older age range.

ELIGIBILITY:
Inclusion Criteria:

* Female and male children with amblyopia age 8-12 years inclusive
* Amblyopic eye visual acuity ≤ 1.0 logMar (20/32-20/200)
* Interocular difference in visual acuity of 0.3 logMAR or more
* Anisometropia or strabismus corrected to <5 pd
* Wearing glasses (if needed) ≥8 weeks
* No longer using standard-of-care treatments for amblyopia
* Informed consent

Exclusion Criteria:

* Prematurity >8 weeks
* Coexisting ocular or systemic disease
* Developmental delay
* History of light-induced epilepsy
* Eye conditions that interfere with eye tracking (nystagmus, wearing RGP contact lenses, paralysis of the extra ocular muscles or any neurological condition that restricts eye movements, ptosis that covers the pupil)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in best-corrected visual acuity of the amblyopic eye compared with baseline best-corrected visual acuity. | 12 weeks
  Change in logMAR best-corrected visual acuity of the amblyopic eye compared with baseline best-corrected visual acuity.

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No